CLINICAL TRIAL: NCT02510924
Title: Role of Airtraq Mobile to Improve Intubation Conditions With Airtraq in Adults With a Simulated Difficult Airway With a Cervical-spine Collar
Brief Title: Role of Airtraq Mobile to Improve Intubation Conditions With Airtraq
Acronym: AirtraqMob
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Patrick Schoettker,MD PD, MD, PD, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 409/14
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Nasal Obstruction; Arthrosis
Keywords: Intubation; Airtraq; General anesthesia; Difficult airway
MeSH Terms: conditions — Nasal Obstruction; Osteoarthritis | interventions — Intubation, Intratracheal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tracheal intubation with Airtraq sp (Active Comparator): Tracheal intubation with Airtraq sp.
  Interventions: Device: Tracheal intubation
- Tracheal intubation with Airtraq Mobile (Experimental): Tracheal intubation with Airtraq Mobile
  Interventions: Device: Tracheal intubation

INTERVENTIONS:
Device: Tracheal intubation — tracheal intubation with Airtraq sp vs Airtraq mobile

SUMMARY:
Airtraq sp has been proven effective for intubating patients presenting with difficult airway.

The Airtraq sp allows visualisation of the tracheal inlet only for the intubator.

By adding a smartphone with a dedicated app (Airtraq Mobile) to the Airtraq sp, the visualisation of the tracheal inlet is possible for all the airway providers.

The investigators aim to demonstrate that the addition of the Airtraq Mobile app improves success rate of intubation (primary endpoint), as well as confort of the airway provider, shortens time for intubation and reduces injury to the patients.

DETAILED DESCRIPTION:
Airtraq sp has been proven effective for intubating patients presenting with difficult airway.

The Airtraq sp allows visualisation of the tracheal inlet only for the intubator.

By adding a smartphone with a dedicated app (Airtraq Mobile) to the Airtraq sp, the visualisation of the tracheal inlet is possible for all the airway providers.

The investigators aim to demonstrate that the addition of the Airtraq Mobile app improves success rate of intubation (primary endpoint), as well as confort of the airway provider, shortens time for intubation and reduces injury to the patients while their neck is imobilized by a cervical collar, creating a simulated difficult airway.

Patients will be included if they necessitate an elective general anesthesia and orotracheal intubation.

Exclusion criteria are related to difficult airway, ASA IV and patient refusal.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia classification 1-3, elective surgey necessitating general anesthesia and intubation, patient consent

Exclusion Criteria:

* American Society of Anesthesia classification 4, patient refusal, history of difficult airway

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-11-05 (Actual); Study Completion 2017-11-05 (Actual)

PRIMARY OUTCOMES:
Success | 180 seconds
  Success of intubation within time frame

SECONDARY OUTCOMES:
Number of attempts | 180 seconds
  Success of intubation within time frame
Number of injuries | 180 seconds
  Injuries within time frame

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schoettker, MD, PD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Dpt of Anesthesiology, University of Lausanne CHUV, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Schoettker P, Corniche J. The AirView Study: Comparison of Intubation Conditions and Ease between the Airtraq-AirView and the King Vision. Biomed Res Int. 2015;2015:284142. doi: 10.1155/2015/284142. Epub 2015 Jun 16. PMID 26161393